CLINICAL TRIAL: NCT03050671
Title: Intermittent Pneumatic Compression in the Lower Limbs: Systemic and Local Effects in Coagulation Status, Microcirculation, Tissue Metabolic Activity and Collagen Production.
Brief Title: Effects of External Leg Compression Devices on Healing and Blood Clotting
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Paul Ackermann, Paul Ackermann M.D, Ph.D., Professor Specialist in Orthopaedic Surgery Orthopaedic Department, Karolinska University Hospital, Karolinska University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: SW2017-01-COAGMET
Record Dates: First submitted 2017-02-09; First posted 2017-02-13 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Venous Stasis; Deep Venous Thrombosis; Healing Wound
MeSH Terms: conditions — Varicose Ulcer; Venous Thrombosis

STUDY DESIGN:
Intervention Model Description: There are two different intervension devices planned to be used in each research subject.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rapid calf-IPC (Active Comparator): Cyclic external compression in both calves through a cuff connected to VenaFlow® Elite System, DJO, CA, USA
  Interventions: Device: Intermittent Pneumatic Compression, Rapid
- subjects under slow calf-IPC (Active Comparator): Cyclic external compression in both calves through a cuff connected to Kendall SCD™ 700, Covidien, Medtronic, USA
  Interventions: Device: Intermittent Pneumatic Compression, Slow

INTERVENTIONS:
Device: Intermittent Pneumatic Compression, Rapid — Cyclic external compression in both calves through a cuff connected to a device which pumps venous blood in a sharp and rapid way
  Arms: Rapid calf-IPC
Device: Intermittent Pneumatic Compression, Slow — Cyclic external compression in both calves through a cuff connected to a device which pumps venous blood in a smooth, slow and progressive way
  Arms: subjects under slow calf-IPC

SUMMARY:
This study aims to compare two different external calf compression devices applied in healthy individuals. These devices are commonly used in medical care in order to prevent the formation of blood clots, for example during immobilization after surgery. We aim to confirm the effects of external cyclic compression on healing and blood clotting and also to identify the one which is more effective.

DETAILED DESCRIPTION:
Aims:

1. To confirm that IPC (intermittent pneumatic compression) has a positive effect on systemic coagulation status, tissue metabolic activity, collagen formation and tissue microcirculation.
2. To compare the above effect of two different IPC devices: one rapid calf-IPC which expels blood from the veins sharp and rapidly and one slow calf-IPC, which pumps the blood in a more gentle and progressive way. This study could also make implications on how the blood flow parameters could be interpreted in the clinical setting, as previous haemodynamic studies have explained the superiority of the rapid device in terms of peak velocity and the superiority of the slow device in terms of total ejected volume per individual stimulus.

Materials and Methods: 10-15 healthy individuals are planned to be recruited. The subjects will be lying in a prone position. A cuff connected with a Calf-IPC device will be wrapped around each calf and will be functioning for 120 minutes. Microdialysis catheters will be inserted with the tips about 1 mm from the volar side of each Achilles tendon. In addition, one adhesive sensor will be applied on each calf just distal to the lower part of the cuff, in order to measure tissue oxygen mixed saturation (INVOS). Blood samples will be taken via a venous catheter in antecubital fossa just before the application of the IPC, and at 30, 60 and 120 minutes. From the serum, several systemic coagulation factors will be measured (tissue plasminogen activator (tPA), plasminogen activator inhibitor type 1 (PAI), tissue factor pathway inhibitor (TFPI), D-dimer, von Willebrand factor and factor VIIa). From the microdialysis diffusate , two groups of substances will be measured: a) metabolites, such as pyruvate and b) collagen macromolecules, such as procollagen type I and III.

The ultimate goal is to assess the role of different IPC patterns on deep venous thrombosis prevention and promotion of tissue healing.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals
* Male gender
* Age 18-60

Exclusion Criteria:

* Smoking
* Severe cardiovascular or renal disease causing pitting oedema
* Previous operation in the lower limbs affecting the vascular or lymphatic system

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only men are being enrolled in order to avoid possible cyclical hormonal influences on blood flow
Enrollment: 10 (Estimated)
Dates: Start 2017-01-18 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
systemic coagulation status | 2 hours
  serum levels of coagulation factors (vWF, tPA, PAI-1, Factor VIIa, TFPI, D-dimer)

SECONDARY OUTCOMES:
local metabolic activity | 2 hours
  Measurement of tissue metabolic products (eg pyruvate) from diffusate extracted with microdialysis in the Achilles paratenon.
collagen production | 2 hours
  Measurement of collagen from diffusate obtained with microdialysis in the Achilles paratenon.
regional microcirculation | 2.5 hours
  Mixed oxygen tissue saturation is continuously measured in the lower leg with infrared spectroscopy

CONTACTS AND LOCATIONS:
Overall Officials: Paul Ackermann, Principal Investigator — Karolinska University Hospital
Locations (1):
- Karolinska university Hospital, Stockholm, Sweden